CLINICAL TRIAL: NCT04276324
Title: Effects of Ten-Weeks Resistance Training on Neuromuscular Performance, Heart Rate Variability, Sleep Quality and Mobility in Persons With Multiple Sclerosis
Brief Title: Effects of Ten-Weeks Power Training on Neuromuscular Performance, Heart Rate Variability, Sleep Quality and Mobility in Persons With Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Jacobo Á. Rubio, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UCAM
Record Dates: First submitted 2020-02-17; First posted 2020-02-19 (Actual); Last update posted 2020-10-23 (Actual); Status verified 2020-10

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Resistance Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Only testing sessions
  Interventions: Other: Testing sessions
- Resistance training group (Experimental): Ten weeks of resistance training
  Interventions: Other: Resistance training; Other: Testing sessions

INTERVENTIONS:
Other: Resistance training — Ten weeks of resistance training
  Arms: Resistance training group
Other: Testing sessions — Testing sessions

SUMMARY:
Multiple Sclerosis (ME) is a degenerative, inflammatory and autoimmune demyelinating disease of the central nervous system, characterized by demyelination due to inflammation and degeneration of the myelin sheaths enveloping nerves of the eye, periventricular grey matter, brain, spinal cord and brainstem. The symptoms associated with MS include symptomatic fatigue, muscle weakness, ataxia, mobility and balance problems or cognitive problems. Strength training has been shown to improve strength and mobility in persons with MS.

ELIGIBILITY:
Inclusion Criteria:

* mild or moderate disability with clinical mild spastic-ataxic gait disorder.
* stable phase of the disease.

Exclusion Criteria:

* Expanded Disability Status Scale (EDSS) < 6.
* relapsing disease within the preceding 12 months.
* corticosteroid treatment within the last months before study inclusion.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2020-03-10 (Actual); Primary Completion 2020-06-15 (Actual); Study Completion 2020-10-15 (Actual)

PRIMARY OUTCOMES:
Maximal Voluntary Isometric Contraction of Knee Extension | Before the program training
Maximal Voluntary Isometric Contraction of Knee Extension | After 10 weeks
Rate of Force Development | Before the program training
Rate of Force Development | After 10 weeks
Central Activation Ratio | Before the program training
Central Activation Ratio | After 10 weeks
Spasticity | Before the program training
  Pendulum test
Spasticity | After 10 weeks
  Pendulum test

SECONDARY OUTCOMES:
Walking speed | Before the program training
  Test 10 m-walks
Walking speed | After 10 weeks
  Test 10 m-walks
Static balance | Before the program training
  Romberg Test with eyes open and closed. Analysis with force plates
Static balance | After 10 weeks
  Romberg Test with eyes open and closed. Analysis with force plates
Functional capacity | Before the program training
  Sit to stand test
Functional capacity | After 10 weeks
  Sit to stand test
Heart Rate Variability | Before the program training
  Sleeping Heart Rate Variability
Heart Rate Variability | After 10 weeks
  Sleeping Heart Rate Variability
Sleep Quality | Before the program training
  Karolinska Sleep Diary and Acelerometry
Sleep Quality | After 10 weeks
  Karolinska Sleep Diary and Acelerometry

CONTACTS AND LOCATIONS:
Overall Officials: Jacobo Á Rubio-Arias, Dr, Principal Investigator — Universidad Católica San Antonio de Murcia
Locations (1):
- Universidad Católica San Antonio, Murcia, Spain

IPD SHARING:
Plan to Share IPD: Yes
The data will be published in a journal
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After the completion of the study